CLINICAL TRIAL: NCT01328587
Title: A Pilot Study of a Thrombopoietin-Receptor Agonist (TPO-R Agonist), Eltrombopag, in Moderate Aplastic Anemia Patients
Brief Title: Eltrombopag for Moderate Aplastic Anemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110134; 11-H-0134
Record Dates: First submitted 2011-04-01; First posted 2011-04-04 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Moderate Aplastic Anemia; Unilineage Bone Marrow Failure Disorders
Keywords: Autoimmunity; Neutropenia; Cytokine; Hematopoiesis; Thrombocytopenia; Aplastic Anemia
MeSH Terms: conditions — Autoimmune Diseases; Neutropenia; Thrombocytopenia; Anemia, Aplastic | interventions — eltrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eltrombopag (Experimental): Eltrombopag will be administered for 16 to 20 weeks at a starting dose of 50mg/day (East Asian ancestry 25mg/day). The dose will decreased and increased (maximum dose 300mg/day) based on safety and response.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag will be administered for 16 to 20 weeks at a starting dose of 150mg/day (East Asian ancestry 75mg /day). The dose will decreased and increased (maximum dose 300mg/day) based on safety and response.

SUMMARY:
Background:

* Moderate aplastic anemia is a blood disease which may require frequent blood and platelet transfusions. Sometimes patients with this disease can be treated with immunosuppressive drugs. Not all patients respond and not all patients are suitable for this treatment.
* Thrombopoietin (TPO) is a protein made by the body. The bone marrow needs TPO to produce platelets. TPO may also be able to stimulate bone marrow stem cells to produce red cells and white cells. However, TPO cannot be given by mouth. This has led researchers to develop the drug eltrombopag, which acts in the same way and can be given by mouth. Eltrombopag has been shown to safely increase platelet numbers in healthy volunteers and in patients with other chronic blood diseases, including severe aplastic anemia. Researchers are interested in looking at whether eltrombopag can be given to people with moderate aplastic anemia and significantly low blood cell counts.

Objectives:

- To evaluate the safety and effectiveness of eltrombopag in people with moderate aplastic anemia or patients with bone marrow failure and unilineage cytopenia who need treatment for significantly low blood cell counts.

Eligibility:

- People at least 2 years of age who have moderate aplastic anemia or bone marrow failure and unilineage cytopenia,and significantly low blood cell counts.

Design:

* Patients will be screened with a physical examination, medical history, blood tests, a bone marrow biopsy, and an eye exam.
* Patients will receive eltrombopag by mouth once a day.
* Patients will have weekly blood tests to monitor the effectiveness of the treatment and adjust the dose in response to possible side effects.
* Patients may continue to take eltrombopag if their platelet count or hemoglobin increases, their requirement for platelet or blood transfusion decreases after 16 to 20 weeks of treatment, and there have been no serious side effects. Access to the drug will continue until the study is closed. Patients will be asked to return for a follow-up visit 6 months after the last dose of medication.

DETAILED DESCRIPTION:
Moderate aplastic anemia (MAA) is a blood disease which can be effectively treated with immunosuppressive drug regimens. However, a significant number of patients have persistent cytopenias. Currently, the treatment of these patients is regular transfusion, which are expensive, inconvenient, and associated with serious side effects related to iron overload, or cytokines such as erythropoietin or G-CSF, which are expensive, and not effective in many patients.

Thrombopoietin (TPO) is a protein made by the body that is important for normal production of platelets by the bone marrow. TPO may also be able to stimulate bone marrow stem cells to produce red cells and white cells. TPO cannot be given by mouth, and as an alternative, a drug, eltrombopag, has been designed that acts in the same way as TPO but is stable and active when given by mouth. Eltrombopag has been shown to safely increase platelet numbers in healthy volunteers and in patients with chronic immune thrombocytopenic purpura (ITP). It has been recently granted accelerated approval by FDA on November 20, 2008 for the treatment of patients with chronic immune thrombocytopenic purpura (ITP) who have had an insufficient response to standard therapies.

We have previously shown encouraging results when eltrombopag is used to treat patients with severe aplastic anemia, with some patients responding with increases in platelets, red cells and white cells. Given these encouraging early preliminary results in our clinical trial using eltrombopag in Severe Aplastic Anemia (SAA), and low toxicity and ease of administration of this drug, we now propose a non-randomized pilot phase II study of eltrombopag in moderate aplastic anemia patients with clinically significant thrombocytopenia or anemia. Patients with MAA may not reach criteria for SAA, but none the less may be transfusion-dependent or have significant symptoms from cytopenias. We hypothesize that patients with MAA as compared to SAA may have a better chance of response, due to better residual marrow function in MAA patients compared to SAA.

Eligible patients can have treated or untreated MAA, as well as counts meeting criteria for MAA following a partial response to treatment with immunosuppression for SAA. We will also include patients with bone marrow failure and unilineage cytopenia. Treatment response for the platelet lineage is defined as platelet count increases to 20,000/microL above baseline at 16 to 20 weeks, or freedom from platelet transfusions for greater than or equal to 8 weeks in transfusion-dependent patients. For patients with anemia (untransfused hemoglobin less than or equal to 8.5 g/dL), a treatment response will be an increase in Hb by greater than or equal to 1.5g/dl at four months, measured on at least 2 serial measurements and sustained for 1 month or more without transfusion support OR for transfusion dependent patients, reduction of units of RCC transfused by 50 percent/8 weeks compared with the pretreatment transfusion number in the previous 8 weeks or transfusion independence (no transfusions for greater than or equal to 8 weeks). Subjects with evidence for a clinical response in any lineage at 16 weeks but not yet meeting full primary endpoint response criteria, and who are tolerating investigational treatment, may receive an additional 4 weeks of eltrombopag and be reassessed after 20 weeks. At that time, if they meet primary endpoint response criteria, they will be eligible to enter the extended access part of the study. If they do not meet primary endpoint response criteria, eltrombopag will be discontinued.

The primary objective is to assess the safety and efficacy of the oral thrombopoietin receptor agonist (TPO-R agonist) eltrombopag in moderate aplastic anemia patients or patients with bone marrow failure and unilineage cytopenia. Secondary objectives include the analysis of the incidence and severity of bleeding, clonal evolution to PNH, clonal chromosomal population in bone marrow, myelodysplasia by morphology, or acute leukemia and the impact on quality of life.

ELIGIBILITY:
* INCLUSION CRITERIA:

Current diagnosis of moderate aplastic anemia or unilineage bone marrow failure disorders.

* Moderate aplastic anemia is defined as aplastic anemia (hypocellular bone marrow for age) with no evidence for other disease processes causing marrow failure, and depression of at least two out of three blood counts below the normal values:

  * ANC less than or equal to 1200/mm(3)
  * platelet count less than or equal to 70,000/mm(3)
  * anemia with hemoglobin less than or equal to 8.5 g/dL and absolute reticulocyte count less than or equal to 60,000/mm(3) in transfusion-dependent patients but not fulfilling the criteria for severe disease defined by depression of two of the three peripheral counts:
  * ANC less than or equal to 500/mm(3)
  * platelet count less than or equal to 20,000/mm(3)
* reticulocyte count less than or equal to 60,000/mm(3)
* Unilineage bone marrow failure disorders are defined:

  * Hemoglobin less than 8.5 g/dL and reticulocyte count less than 60,000 or red cell transfusion dependent and hypocellular to normocellular bone marrow for age with significantly reduced erythroid precursors.
  * OR thrombocytopenia less than or equal to 30,000/uL or platelet transfusion dependent and hypocellular to normocellular bone marrow for age with reduced megakaryocytes.
* No evidence of viral or drug suppression of the marrow, dysplasia, or underproduction anemias secondary to B12, folate, iron or other reversible causes.

Platelet transfusion dependent is defined as the need for platelet transfusion due to platelet counts of < 10,000/microL with no bleeding (prophylactic transfusion) or < 20,000/microL with bleeding (therapeutic transfusion). Red cell transfusion dependent is defined as transfusion of greater than 4 units of blood in the 8 weeks prior to study entry.

Age greater than or equal to 2 years old

Weight greater than 12 kg

EXCLUSION CRITERIA:

Known diagnosis of Fanconi anemia

Counts that meet criteria for severe aplastic anemia

Infection not adequately responding to appropriate therapy

HIV positivity

Creatinine > 2.5 mg/dL

Bilirubin > 2.0 mg/dL, including congenital abnormalities in the bilirubin count

SGOT or SGPT >5 times the upper limit of normal

Hypersensitivity to eltrombopag or its components

Female subjects who are nursing or pregnant or are unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential

Evidence of an active malignant hematological or clonal disorder, or abnormal cytogenetic studies of the bone marrow performed within 12 weeks of study entry.

Unable to understand the investigational nature of the study or give informed consent or does not have a legally authorized representative or surrogate that can provide informed consent

Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient's ability to tolerate protocol therapy, or that death within 7-10 days is likely.

Treatment with horse or rabbit ATG or Campath within 6 months of study entry.

Treatment with cytokines such as G-CSF or Erythropoietin.

Subjects with known cirrhosis in severity that would preclude tolerability of eltrombopag as evidenced by albumin less than 35g/L.

Life expectancy of less than 3 months

Patients with an active diagnosis of cancer who have received chemotherapeutic treatment or other specific antineoplastic drugs or radiation therapy within 6 months of study entry.

Unable to take investigational drug

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-04-01; Primary Completion 2018-03-30 (Actual); Study Completion 2025-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia E Dunbar, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Young NS, Barrett AJ. The treatment of severe acquired aplastic anemia. Blood. 1995 Jun 15;85(12):3367-77. No abstract available. PMID 7780125
- [Background] Young NS, Calado RT, Scheinberg P. Current concepts in the pathophysiology and treatment of aplastic anemia. Blood. 2006 Oct 15;108(8):2509-19. doi: 10.1182/blood-2006-03-010777. Epub 2006 Jun 15. PMID 16778145
- [Background] Zeng W, Maciejewski JP, Chen G, Risitano AM, Kirby M, Kajigaya S, Young NS. Selective reduction of natural killer T cells in the bone marrow of aplastic anaemia. Br J Haematol. 2002 Dec;119(3):803-9. doi: 10.1046/j.1365-2141.2002.03875.x. PMID 12437663
- [Derived] Fan X, Desmond R, Winkler T, Young DJ, Dumitriu B, Townsley DM, Gutierrez-Rodrigues F, Lotter J, Valdez J, Sellers SE, Barranta ME, Shalhoub RN, Wu CO, Albitar M, Calvo KR, Young NS, Dunbar CE. Eltrombopag for patients with moderate aplastic anemia or uni-lineage cytopenias. Blood Adv. 2020 Apr 28;4(8):1700-1710. doi: 10.1182/bloodadvances.2020001657. PMID 32330244
- [Derived] Giudice V, Wu Z, Kajigaya S, Fernandez Ibanez MDP, Rios O, Cheung F, Ito S, Young NS. Circulating S100A8 and S100A9 protein levels in plasma of patients with acquired aplastic anemia and myelodysplastic syndromes. Cytokine. 2019 Jan;113:462-465. doi: 10.1016/j.cyto.2018.06.025. Epub 2018 Jun 27. PMID 29958797
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-H-0134.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Eltrombopag: Patients will receive Eltrombopag ( thrombopoietin receptor agonist) by mouth once a day.
Period: Overall Study
Arm/Group | Eltrombopag
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 27
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 23
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Drug Responders
Description: Defined by changes in platelet count and/or platelet transfusion requirements or hemoglobin (Hb) and/or PRBC transfusion requirements and the toxicity profile as measured by CTCAE. Response for platelet lineage is defined as absolute increase of ≥20x10^9/L above baseline at 16 or 20 weeks, with at least 2 serial measurements performed 1 week apart and sustained for 1 month or more without platelet transfusions, or for transfusion dependent patients stable platelet counts with transfusion independence for ≥ 8 weeks. Patients with anemia (untransfused hemoglobin ≤ 8.5 g/dL), a response will be an increase in Hb by ≥1.5g/dL at 4 months, with at least 2 serial measurments and sustained for 1 month or more without transfusion support OR for transfusion dependent patients, reduction of units of RCC transfused by 50%/8 weeks compared with the pretreatment transfusion number in the pretreatment transfusion number in the previous 8 weeks or transfusion independence (no transfusions ≥ 8 weeks).
Time Frame: 16-20 weeks from start of drug
Measure: Count of Participants; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 34
Participants | 17

ADVERSE EVENTS:
Time Frame: 42 months from enrollment
Arm/Group | Eltrombopag
All-Cause Mortality (participants affected / at risk) | 1/34
Serious Adverse Events (participants affected / at risk) | 1/34
Other Adverse Events (participants affected / at risk) | 29/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=34)
Metastatic Ovarian CA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=34)
blood and lymphatic system d/s other, specify (Blood and lymphatic system disorders) | 1
Gingival Bleeding (Blood and lymphatic system disorders) | 1
Hematuria (Blood and lymphatic system disorders) | 1
spleen disorder/splenic varices (Blood and lymphatic system disorders) | 1
spleen disorder/splenomegaly (Blood and lymphatic system disorders) | 1
abdominal edema (Cardiac disorders) | 1
BLE edema (Cardiac disorders) | 1
dyspnea on exertion (Cardiac disorders) | 1
fatigue (Cardiac disorders) | 2
fatigue/angina (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
scrotal edema (Cardiac disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
External Ear pain/discomfort (Ear and labyrinth disorders) | 1
otitis media/external ear inflammation (Ear and labyrinth disorders) | 1
Burning Eyes (Eye disorders) | 1
eye tingling/pain (Eye disorders) | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Blood in stool (Gastrointestinal disorders) | 1
collagenous colitis (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
diarrhea (Gastrointestinal disorders) | 6
diarrhea/stomach cramps (Gastrointestinal disorders) | 1
epigastric tenderness (Gastrointestinal disorders) | 1
food poisoning (Gastrointestinal disorders) | 1
foodpoisoning/gastroenteritis (Gastrointestinal disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
GI illness(nausea, vmitting, diarrhea) (Gastrointestinal disorders) | 1
Gi symptoms (Gastrointestinal disorders) | 1
Gum Bleeding (Gastrointestinal disorders) | 1
h pylori (Gastrointestinal disorders) | 1
intermittent lower pelvic pain (Gastrointestinal disorders) | 1
Loose Stool (Gastrointestinal disorders) | 1
Loose stools (Gastrointestinal disorders) | 2
Mild constipation (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 6
nausea/diarrhea (Gastrointestinal disorders) | 1
nausea/vomiting (Gastrointestinal disorders) | 2
nausea/vomiting/abd cramps (Gastrointestinal disorders) | 1
Pinworms (Gastrointestinal disorders) | 1
rectal bleeding (Gastrointestinal disorders) | 1
Viral Gastroenteritis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Worsening GERD (Gastrointestinal disorders) | 1
chills (General disorders) | 1
facial edema (General disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 3
Flu like symptoms (General disorders) | 1
Headache (General disorders) | 4
Influenza (General disorders) | 1
intermittent night sweats (General disorders) | 1
LE edema (General disorders) | 1
lightheaded (General disorders) | 1
cirrhosis (Hepatobiliary disorders) | 1
Elevated AST (Hepatobiliary disorders) | 1
Elevated Bilirubin (Hepatobiliary disorders) | 1
portal hypertension (Hepatobiliary disorders) | 1
CTLA 4 deficiency (Immune system disorders) | 1
Abscessed Tooth (Infections and infestations) | 2
C diff (Infections and infestations) | 1
strep throat (Infections and infestations) | 1
tooth #30 infection (Infections and infestations) | 1
UTI (Infections and infestations) | 1
UTI/Inflammed prostate (Infections and infestations) | 1
yeast infection (Infections and infestations) | 1
easy bruising (Injury, poisoning and procedural complications) | 1
Foot pain from fall (Injury, poisoning and procedural complications) | 1
shoulder pain from fall (Injury, poisoning and procedural complications) | 1
ALT increase (Investigations) | 1
AST increase (Investigations) | 1
Elevated Liver Enzymes (Investigations) | 1
yellowing skin/eye (Investigations) | 1
muscle cramps (Musculoskeletal and connective tissue disorders) | 1
R Breast Pain (Musculoskeletal and connective tissue disorders) | 1
R Calf Cramps (Musculoskeletal and connective tissue disorders) | 1
Rib pain (Musculoskeletal and connective tissue disorders) | 1
dizzy (Nervous system disorders) | 1
fingers tingly'-peripheral sensory neuropathy (Nervous system disorders) | 1
headaches (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Dark urine (Renal and urinary disorders) | 1
UTI (Renal and urinary disorders) | 2
Chest cold (Respiratory, thoracic and mediastinal disorders) | 1
Cold Sxs (Respiratory, thoracic and mediastinal disorders) | 2
cough (Respiratory, thoracic and mediastinal disorders) | 1
dry cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea on Exertion (Respiratory, thoracic and mediastinal disorders) | 1
Flu-like symptoms (Respiratory, thoracic and mediastinal disorders) | 1
hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Mild Flu-like symptoms (Respiratory, thoracic and mediastinal disorders) | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
sinus pressure (Respiratory, thoracic and mediastinal disorders) | 1
sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1
sore throat (Respiratory, thoracic and mediastinal disorders) | 1
URI (Respiratory, thoracic and mediastinal disorders) | 4
Viral URI (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
facial rash (Skin and subcutaneous tissue disorders) | 1
left post auricular skin (Skin and subcutaneous tissue disorders) | 1
Rash on Arm (Skin and subcutaneous tissue disorders) | 1
Shingles (Skin and subcutaneous tissue disorders) | 1
skin rash (Skin and subcutaneous tissue disorders) | 1
vitiligo (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT01328587/Prot_SAP_000.pdf